CLINICAL TRIAL: NCT01334450
Title: Deep-TMS for the Treatment of Alzheimer Disease Patients
Brief Title: Transcranial Magnetic Stimulation (TMS) Treatment for Alzheimer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Meiner Ze'ev, Hadassah Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0316
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2011-04

CONDITIONS: Alzheimer Disease
Keywords: Improvement of ADAS-COG
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Frequency TMS to prefrontal cortex (Active Comparator)
  Interventions: Device: TMS , H2-coil
- Low Frequency TMS to Prefrontal cortex (Active Comparator)
  Interventions: Device: TMS , H2-coil
- Sham TMS on Prefrontal Cortex (Sham Comparator)
  Interventions: Device: TMS , H2-coil

INTERVENTIONS:
Device: TMS , H2-coil — Trans cranial magnetic stimulation with H2-coil
  Other Names: Not relevant

SUMMARY:
Transcranial Magnetic Stimulation (TMS) for treatment of Alzheimer disease.

DETAILED DESCRIPTION:
Transcranial Magnetic Stimulation (TMS) for treatment of Alzheimer disease.

Alzheimer's disease (AD) is the leading cause of dementia and cognitive deteriorating in the advanced age. The current medical treatment of AD is mainly symptomatic and has many limitation. This main target of this study is to determine the safety and efficacy of transcranial magnetic stimulation (TMS) using novel coil design (H2) for stimulation of deep brain structures concomitantly with regular treatment in Alzheimer's disease (AD) patients. TMS acts by generating magnetic fields in the brain which simulate neuro-chemical changes and stimulate neuronal activity translating into increased secretion of growth factors such as brain derived neurotrophic factor (BDNF). Hence it is postulated that TMS will have a positive effect on the cognitive and behavioral symptoms of patients with AD and may ameliorated the progression of the disease. The treatment is non-invasive, with no significant side effects, and no need of hospitalization or anesthesia. The trial is phase IIb double blind study including 45 AD patients ages between 50 to 80 with mild or moderate AD (Mini Mental State Examination [MMSE] between 16 to 26) divided into 3 groups. All participants will receive standard medical therapy for AD. In addition, patients recruited for the study will receive 16 sessions of TMS with the H2 coil over 8 weeks. The first group will receive excitatory stimulation of 10 Hz over the prefrontal and parietal cortex, the second group will receive inhibitory stimulation of 1 Hz over similar brain areas and control patients will receive the same amount of Sham sessions. Patient will receive 3 treatments per week in the first 3 weeks and than 1 treatment per week for additional 4 weeks. Patients will be evaluated before the treatments, after 8 weeks of treatment and after another 8 weeks without treatment. The evaluations will include cognitive function according to ADAS-COG and MMSE, Activity of daily living (ADL) functions according to ADSC-ADL, behavioral function according to the Neuropsychiatric Inventory (NPI), depression according to the Cornell Scale for Depression in Dementia (CSDD), care giver satisfaction according to the RUD LITE scale and computerized cognitive evaluation according to the NEXING battery. We expect that the cognitive, behavioral and ADL functions will improve better in the study group as compared to the Sham treated group. From previous trial of TMS in neurological patients, although not in AD, we anticipate that adverse events rate will be similar between groups proving the safety of deep TMS treatment in patients with AD. In case our hypothesis will be proven, deep TMS treatment will be added as an important modality to the conventional therapy of AD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 50-85.
2. Diagnosed with Alzheimer's disease for at least half a year (by the DSM-IV criteria).
3. Scored between 16-26 on the MMSE.
4. Received drug therapy for their disease, with each treatment having been administered at an acceptable dosage for at least 5 weeks.
5. Existence of a routine therapist for changes or adverse effects reports.
6. Existence of Alzheimer diagnosis by CT or MRI tests.
7. Answered in the negative to all questions in the pre-TMS treatment safety questionnaire.
8. Gave their oral and written consent to participate in the trial.

Exclusion Criteria:

1. An additional neurological disorder.
2. Severe psychiatric disorder.
3. Uncontrolled hypertension, beyond 170/110.
4. History of epilepsy, seizure, or heat convulsion or History of epilepsy or seizure in first degree relatives.
5. History of head injury or stroke.
6. History of metal implants in the head (except dental fillings)or History of surgery entailing metallic implants or known history of any metallic particles in the eye, implanted cardiac pacemaker, cochlear implants, use of neurostimulators, or any medical pumps.
7. History of migraines in the last six months.
8. History of drug or alcohol abuse.
9. Inadequate communication with examiner.
10. Participation in another clinical study, either concurrent with this trial or in the 3 months preceding it.
11. Inability to sign a consent form.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
cognitive functioning score by ADAS-COG | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Meiner, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem District, Israel, Israel